CLINICAL TRIAL: NCT03148730
Title: Manual vs Automated Optimization of Anesthesia, Analgesia, Fluid Management and Ventilation Using Closed-loop Systems: Impact On The Incidence Of POCD In Elderly Patients Undergoing Moderate to High Risk Surgery
Brief Title: Manual vs Automated Anesthesia : Impact On The Incidence Of POCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P2015/539 / B406201526591
Record Dates: First submitted 2017-05-01; First posted 2017-05-11 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: 2 groups one = manually conducted anesthesia second = fully automated anesthesia, analgesia, ventilation and fluid management
Who Masked: Participant, Outcomes Assessor
Masking Description: single blinded ( outcome assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual group (No Intervention): This group will have a standard of care anesthesia. All the drugs, fluid and adjustement of ventilation settings will be done manually by the supervising anesthesiologist using the same drugs and fluids as the closed-loop group
- automated closed-loop group (Experimental): This group will have a fully automated anesthesia, analgesia , ventilation and fluid management using 3 indenpendent closed-loop systems same drugs used in both groups ( propofol and remifentanil, Plasmalyte and /or Voluven)
  Interventions: Device: closed-loop group

INTERVENTIONS:
Device: closed-loop group — Use of 3 indenpendent closed-loop systems to deliver the propofol, remifentanil, fluid and to adjust ventilation
  Arms: automated closed-loop group

SUMMARY:
This study will be the first study to report the combined use of three independent closed-loop systems together to assist clinicians in titrating anesthesia, analgesia, fluid and optimize ventilation in frailty old patients undergoing moderate to high risk surgery. The potential benefits of optimizing the control of these variables by advanced closed loop systems are two-fold. Firstly, this will likely decrease the variance of delivered care and reduce deviation from the established standards, resulting in improved post operative cognitive outcomes in elderly patients. Secondly, this would establish a precedent that automated intraoperative systems have strong clinical significance and are more than "complicated toys", which is unfortunately how they are perceived now.

Hypothesis: Automated control of anesthetic depth (minimal episodes of overly deep or light anesthesia) and hemodynamics (via improved volume administration) can decrease the occurrence of postoperative cognitive dysfunction in elderly patients undergoing moderate to high risk surgery (Better MOCA test in the postoperative period compared to the manual group [+ two points in average])

DETAILED DESCRIPTION:
Elderly patients comprise more than 40% of all surgical patients in the USA per year and generate an even larger proportion of total healthcare costs with a sizable amount occurring during the postoperative period 1.. Therefore, reducing postoperative morbidity and mortality is a major concern in clinical practice and medical research moving forward. Cognitive dysfunction and dependence on caregivers represents two major risk factors in the elderly, especially following general anesthesia. The current literature indicates that POCD results in a mortality rate of 10% at 6 months for patients at least 70 years old and causes loss of functional capacity in an additional 20%. Overall, this results in an approximately 1 of 3 patients experiencing a negative cognitive impact following general anesthesia without optimization of anesthetic depth. In this context, continuous monitoring of the depth of anesthesia using a bispectral index (BIS) sensor may reduce the occurrence of postoperative impairments by via improved control of the anesthetic depth, especially over-sedation.

Despite steady improvements in surgical safety throughout recent years, the application of perioperative therapies still has the potential to be improved, especially regarding compliance to evidence-based recommendations.2, 3 Specifically, simply being surrounded by established monitors does not ensure that proper therapies are delivered most effectively or consistently to all patients - there must also be appropriate and timely interventions. Concordantly, large variations in patient care still exist and have been correlated with large variations in patient outcomes.4 Looking at the safety record that automation has achieved in fields ranging from manufacturing to commercial flight, medical researchers have developed devices utilizing self-contained feedback technologies (CLS) in an attempt to decrease the variability in treatment delivery with the ultimate goal of improving patient care. This development has flourished within anesthesiology, mainly via physiological closed-loop controlled devices. These systems are able to automatically adjust a therapeutic intervention based on continuous feedback from various physiological sensors.5 The best described systems have been closed-loop delivery of anesthetics, analgesics,6-11 volatile agents, insulin, and most recently, fluids 5, 12-14 and vasopressors.15-17 Overall, these systems have been shown to improve the consistency of intervention when compared to manual administration.10, 18, 19 Additionally, computer-assistance for clinical care will allow anesthesia providers to increase their accuracy and consistency, improve their awareness, and allow them to instead focus on more complex tasks.

Over the past years, members of our group have developed a dual closed-loop controller allowing the automated titration of propofol and remifentanil guided by the bispectral index (BIS).11, 20-22 The investigators also have created an adaptative closed-loop system for fluid titration using goal directed fluid therapy (GDFT) strategies guided by a minimally invasive cardiac output monitor.5 The investigator has previously demonstrated the superiority of a controller versus human-guided anesthesia in maintaining a target of BIS between 40 and 60 while limiting the incidence of overly deep anesthesia, which is often associated with the occurrence of a cognitive dysfunction in the elderly 23 Very recently, the principal investigator submitted research evaluating the simultaneous use of 2 closed-loop system (anesthesia, analgesia and fluid management) in a pilot study of high risk vascular patients.

Objectives: The main objective of this prospective randomized single-blinded controlled study is to compare manual versus automated administration of anesthesia, analgesia, fluid and ventilation with regard to the incidence of postoperative cognitive dysfunction (POCD) in elderly patients undergoing high risk surgery. POCD will be assessed by a psychiatrist and/or a psychologist preoperatively, on postoperative day 3-10 (depending on the type of surgery) and at 3-months postoperatively. Additionally, quality of life and quality of recovery will also be self-assessed before surgery, before hospital discharge and at 3 month post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > or equal 60 years old
* ASA score I-III
* Scheduled for non cardiac surgery under total intravenous anesthesia
* Self sufficient (living at home or in non medical institution)
* MOCA test preop > 23/30
* No Stroke, alzeihmer, Parkinson disease
* Written informed consent signed

Exclusion Criteria:

* Allergy to propofol or remifentanil
* MOCA test < 23/30
* Visual or hearing deficiency
* Atrial fibrillation, or other Contra indication to the use of dynamic parameters of fluid responsiveness.
* Chronic renal failure ( creatinin level maximum at 2 mg/ml; no dialysis)
* Large liver resection : our center has a strict fluid /CVP fluid restriction in place

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative cognitive dysfunction (POCD) | first month
  assessment of the POCD using the MOCA test ( done by a psychiatrist and a psychologist). This will be done preoperatively, at postoperative day 3-5 for moderate risk surgery and postoperative day 7-10 for high risk surgery

SECONDARY OUTCOMES:
Assesment of the incidence of POCD using different others tests: | Before Surgery
  1) assessment of verbal episodic memory (van der linden et al, 2004: RL/RI-16 2) Digit Span (assessment of short term memory: in order and reverse order (assessment of working memory) 3) Stroop test: assessment of inhibition (Chatelois, 1993). This will be done day the before surgery
Assesment of the incidence of POCD using different others tests: | day 5 after surgery
  1) assessment of verbal episodic memory (van der linden et al, 2004: RL/RI-16 2) Digit Span (assessment of short term memory: in order and reverse order (assessment of working memory) 3) Stroop test: assessment of inhibition (Chatelois, 1993). This will be done on postoperative day 3-5 (for moderate risk surgery)
Assesment of the incidence of POCD using different others tests: | day 10 after surgery
  1) assessment of verbal episodic memory (van der linden et al, 2004: RL/RI-16 2) Digit Span (assessment of short term memory: in order and reverse order (assessment of working memory) 3) Stroop test: assessment of inhibition (Chatelois, 1993). This will be done on postoperative day 7-10 for high risk surgery
Long term incidence of POCD | month 3 post surgery
  results of the MOCA test
Assessment of the Quality of life EQ-5D-5L | 3 months
  self assessment by the patient: done the day before surgery and at month 3 post surgery
Assessment of Quality of recovery (QoR) | first month
  self assessment by the patient: QoR-15 items: questionnaire done before surgery to provide baseline data and then repeated after surgery (post operative day 3 for moderate risk surgery and postoperative day 7for high risk surgery).
Amount of i.v drugs used ( propofol, remifentanil, vasopressors) | first 24 hours
  amount of iv drugs used during the surgery
Amount of total fluid infused to the patient | first 24 hours
  comparison of the amount of fluid administered to the patients between groups
Mean BIS values and Burst suppression ratio (BSR) incidence defined as a period of isoelectric cortical signal with a treshold at 10% for > 1 minutes. | first 24 hours
  comparison of the mean BIS values and occurrence of BSR between groups
mean arterial pressure (MAP) during surgery | first 24 hours
  comparison of the mean values of these variables between both groups
Mean : mean stroke volume, stroke volume variation and cardiac output and cardiac index | first 24 hours
  comparison of the mean values of these variables between both groups
Incidence of postoperative complications (major and minor) | From date of surgery until day 30 after surgery
  comparison of the incidence of postoperative complications between both groups
Length of stay in the intensive care unit (ICU) and/or postanesthesia care unit (PACU) | From date of surgery until the date of Postanesthesia or intensive care setting discharge or date of death from any cause assessed up to 100 weeks after surgery
  comparison of the length of stay between both groups
Length of stay in the hospital ( | From date of surgery until the date of hopital discharge or date of death from any cause assessed up to 100 weeks after surgery
  comparison of the hospital length of stay between both groups
Mortality at day 30 | 30 days
  death at 1 month
Mortality at month 3 | 3 months
  death at 3 months
Comparison of performance of the automated system vs the manual group | first 24 hours
  defined as the time of the surgery spent with a BIS values [40-60] and a SVV <13% and/or a CI > 2.5 l/min/m2 for
Occurrence of arterial hypotension (mean arterial pressure (MAP) < 65 mmHg) | first 24 hours
  MAP < 65 mmHg
Occurrence of awarness | first 24 hours
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Joosten, M.D, Principal Investigator — Erasme
Locations (1):
- Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided